CLINICAL TRIAL: NCT03818555
Title: A Prospective, Multicenter, Postmarket Study of Sebacia Microparticles Treatment in Patients Using Topical Acne Products for Mild to Moderate Inflammatory Acne Vulgaris
Brief Title: Sebacia Postmarket Study of Real-World Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sebacia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SEB-0550
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Sebacia Microparticles Treatment (Other)
  Interventions: Other: Sebacia Microparticles Treatment

INTERVENTIONS:
Other: Sebacia Microparticles Treatment — Sebacia Microparticles procedure involving microparticles and 1064 nm laser. Three treatment procedures over a two-week period.
  Other Names: Sebacia treatment, Microparticles and Nd:Yag laser treatment

SUMMARY:
Postmarket study of Sebacia Microparticles treatment during adoption into clinical use for patients with mild to moderate inflammatory acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate facial inflammatory acne vulgaris (IGA 2 or 3)
* Between 10 and 50 papules/pustules
* Fitzpatrick skin phototype I, II or III
* Able to provide informed consent and comply with study schedule and other requirements

Exclusion Criteria:

* Moderately severe or severe acne vulgaris (IGA 4 or 5)
* Nodulocystic acne, significant scarring or excoriation
* Requires oral retinoid, antibiotic or corticosteroid for acne
* New or fluctuating hormone or hormone-regulating therapy
* Photosensitivity or allergy to gold
* Medical or mental health condition that would pose a risk to patient or impair treatment and evaluation

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 125 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Inflammatory Lesion Count | Months 2, 3, 6, 9 and 12
  Percent change in number of inflammatory lesions from baseline

SECONDARY OUTCOMES:
Investigator's Global Assessment | Months 2, 3, 6, 9 and 12
  Percent of subjects clear (IGA 0) or almost clear (IGA 1)
Physician's Overall Assessment of Improvement | Months 2, 3, 6, 9 and 12
  Categorical improvement from baseline (worse, no change, minimal, moderate, marked, complete)

CONTACTS AND LOCATIONS:
Overall Officials: VP, Clinical & Regulatory Affairs, Study Director — Sebacia, Inc.
Locations (6):
- United States (6):
  - Miami Dermatology & Laser Institute, Miami, Florida
  - Dermatology Institute of Boston, Boston, Massachusetts
  - International Clinical Research, Murfreesboro, Tennessee
  - Austin Institute for Clinical Research - Central, Austin, Texas
  - Austin Institute for Clinical Research - Pflugerville, Pflugerville, Texas
  - Premier Clinical Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Company Website — http://www.sebacia.com